CLINICAL TRIAL: NCT03780023
Title: Pilot Study to Measure the Health-related Quality of Life Associated With a Physician Communication Intervention for Prostate Cancer Patients Undergoing Definitive or Post-operative Radiation Treatment.
Brief Title: CCRO044: Quality of Life Assessments Associated With a Physician Communication Intervention for Prostate Cancer Patients
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 1072827
Record Dates: First submitted 2018-12-06; First posted 2018-12-19 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Prostate Adenocarcinoma
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — All patients will receive three questionnaires at four different time points during their radiation treatment. The time points are 1) before treatment, 2) during the first week of treatment, 3) at the end of treatment (6-8 weeks after treatment begins), and 4) one year after treatment ends.

SUMMARY:
A generic cancer health-related quality of life measure will be used to assess the impact of the patient-specific radiation therapy plan review using the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)-C30. Patient psychosocial adjustment will be assessed by the Memorial Anxiety Scale for prostate cancer and the EORTC QLQ-C30 subdomain. Physician communication will be assessed with the UC Davis Physician Communication adapted from the Cologne Patient Questionnaire.

The study will characterize the above health-related quality of life (HRQL) scores (EORTC QLQ C-30, the Memorial Anxiety Scale, and the UC Davis Physician Communication) prior to initiation of radiation (baseline), during the first week of treatment, at the end of radiation treatment (6-8 weeks following initiation of treatment), and 12 months after treatment ends.

DETAILED DESCRIPTION:
The primary purpose of this pilot study is to assess the feasibility of administrating a battery of HRQL measures after the planned intervention is administered. Because distributional information on the proposed HRQL measure has not been previously collected in prostate cancer patients, this pilot study will provide the necessary descriptive statistical information for the planned endpoint measures (summary scores for the HRQL battery) to help plan a randomized trial evaluating the efficacy of the patient-provider communication intervention. Men who are receiving definitive or post-operative radiation therapy for management of prostate cancer at the University of California (UC) Davis will be recruited.

The study will administer a validated quality of life instrument (EORTC QLQ-C30), a previously validated psychosocial instrument (Memorial Anxiety Scale), and assessment of physician-patient communication using a new UC Davis Physician Communication Assessment adapted from the validated Cologne Patient Questionnaire. The study will administer these questionnaires prior to initiation of radiation (baseline), during the first week of treatment, at the end of radiation treatment (6-8 weeks following initiation of treatment), and 12 months after treatment ends.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of prostate adenocarcinoma over the age of 18 years
2. Low, intermediate or high risk as defined by D'Amico risk groups treated with dose escalated conventional fractionated radiation therapy
3. Patient deemed clinically appropriate for definitive, adjuvant or salvage radiation.
4. Patient most provide study specific informed consent prior to study entry.
5. Androgen deprivation allowed
6. Pelvic lymph radiation therapy allowed for high risk disease

Exclusion Criteria:

1. Metastatic prostate cancer
2. Positive pelvic nodes
3. Patients treated with radiation for palliative intent
4. Prior radiation therapy to the pelvis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This is a prostate cancer protocol.
Study Population: Men age 18 and over with a diagnosis of prostate adenocarcinoma that is not characterized by metastatic cancer or positive pelvic nodes.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Change in health-related quality of life | Baseline, 6 to 8 weeks
  The mean change in scores on the EORTC QLQ-C30 scale from pre-treatment to post-treatment. This scale has functional, global health, and symptoms subscales/items all scored from 0 to 100. Higher scores on these subscales indicate high level of functioning, high quality of life, and high level of symptomatology, respectively.
Change in psychosocial health | Baseline, 6 to 8 weeks
  The mean change in scores on the Modified 18-item Memorial Anxiety Scale for Prostate Cancer from pre-treatment to post-treatment. The scale consists of 18 items (e.g. "I thought about prostate cancer even though I didn't mean to.") scored on a scale from 0 ("not at all") to 3 ("often"). Total scores range from 0 to 54, with higher scores indicating higher levels of anxiety.
Change in physician-patient communication | Baseline, 6 to 8 weeks
  The mean change in scores on the UC Davis Physician Communication Assessment from pre-treatment to post-treatment. This scale was adapted from the validated Cologne Patient Questionnaire, which has subscales measuring devotion, support, information, and shared decision-making. Participants indicate their level of agreement with each item, from "totally disagree" to "totally agree."

CONTACTS AND LOCATIONS:
Overall Officials: Richard K Valicenti, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided